CLINICAL TRIAL: NCT05458089
Title: 18F-FDG PET/CT in the Diagnosis of Tuberculous Pericarditis
Status: Completed | Type: Observational
Sponsor: Wuxi No. 4 People's Hospital (Other)
Responsible Party: Principal Investigator, Chunjing Yu, director of the nuclear medicine, Wuxi No. 4 People's Hospital
Other Study IDs: Wuxi4PH-2022-01
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Diagnostic Self Evaluation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- tuberculous pericarditis with 18F-FDG uptake: patients confirmed with tuberculous pericarditis presenting 18F-FDG uptake
  Interventions: Diagnostic Test: 18F-FDG
- tuberculous pericarditis without 18F-FDG uptake: patients confirmed with tuberculous pericarditis presenting no 18F-FDG uptake
  Interventions: Diagnostic Test: 18F-FDG

INTERVENTIONS:
Diagnostic Test: 18F-FDG — 18F-FDG intravenous injection

SUMMARY:
A total of 11 patients confirmed with tuberculous pericarditis were enrolled in this study to analyze the diagnostic value of 18F-FDG PET/CT for tuberculous pericarditis.

DETAILED DESCRIPTION:
A total of 11 patients with tuberculous pericarditis, who underwent 18F-FDG PET/CT from January 2015 to February 2022 in the affiliated hospital of Jiangnan university were retrospectively reviewed in this study to analyze the diagnostic value of 18F-FDG PET/CT in tuberculous pericarditis.

ELIGIBILITY:
Inclusion Criteria:

patients confirmed as tuberculous pericarditis through follow-up.

Exclusion Criteria:

patients confirmed as other pericarditis through follow-up.

Ages: 48 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 11 patients confirmed with tuberculous pericarditis were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
the diagnostic sensitivity of 18F-FDG PET/CT for tuberculous pericarditis | 01,2015-02,2022
  the diagnostic sensitivity of 18F-FDG PET/CT for tuberculous pericarditis

IPD SHARING:
Plan to Share IPD: No